CLINICAL TRIAL: NCT00683176
Title: Effect of Choline Fenofibrate (SLV348) on Macular Edema Measured by Optical Coherence Tomography in Subjects With Diabetic Macular Edema - a One-year, Placebo-Controlled, Randomized Study
Brief Title: Effect of Choline Fenofibrate (SLV348) on Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Products (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S348.2.001; 2008-001064-37 (EudraCT Number)
Record Dates: First submitted 2008-05-16; First posted 2008-05-23 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; OCT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Choline Fenofibrate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline Fenofibrate — 135 mg
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of choline fenofibrate on the regression of macular edema in eyes of subjects with type 2 diabetes mellitus (T2DM) presenting with diabetic macular edema (DME)

ELIGIBILITY:
Inclusion Criteria

* With DME in at least one eye of the subject and this eye presenting with macula thickness ≥ 300 µm on OCT examination at baseline in at least one of the 5 following zones: center zone, or superior inner zone, or nasal inner zone, or inferior inner zone, or temporal inner zone, confirmed after central reading of the OCT;
* When laser treatment can be safely postponed by up to at least 3 months;
* With established T2DM and HbA1c < 10%;
* With systolic blood pressure (SBP) or diastolic blood pressure (DBP) < 160/90 mmHg;
* With documented elevated triglyceride levels (TG >=150 mg/dL [1.70 mmol/L]) at the screening visit or in the previous 3 months.

Exclusion Criteria

* Previous laser photocoagulation;
* Eye retinal thickening results from epiretinal membranes or vitreomacular traction; glaucoma;
* Poor visual acuity: visual acuity of 20/800

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Total macular volume measurement on OCT, after central reading (assessed at baseline and after 3, 6, 9 and 12 months of treatment) | 12 months

SECONDARY OUTCOMES:
OCT variables (Retinal Thickness, Retinal thickening) | 12 months
ETDRS macular and hard exudate grading, E-ETDRS visual acuity, ETDRS retina grading, at least 2 step progression, Laser photocoagulation for diabetic macular edema | 12 months
Lipids | 12 months
SBP/DBP, Urinary albumin excretion rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jean-Claude Ansquer, MD, Study Director — Abbott Products
Locations (21):
- Bulgaria (4):
  - Site Reference ID/Investigator# 54268, Sofia
  - Site Reference ID/Investigator# 54291, Sofia
  - Site Reference ID/Investigator# 54279, Sofia
  - Site Reference ID/Investigator# 54273, Sofia
- Czechia (4):
  - Site Reference ID/Investigator# 54267, Brno
  - Site Reference ID/Investigator# 54282, Ostrava-Vitkovice
  - Site Reference ID/Investigator# 54283, Prague
  - Site Reference ID/Investigator# 54270, Ústí nad Labem
- Site Reference ID/Investigator# 54274, Glostrup Municipality, Denmark
- Germany (2):
  - Site Reference ID/Investigator# 54263, Leipzig
  - Site Reference ID/Investigator# 54284, Münster
- Hungary (3):
  - Site Reference ID/Investigator# 54269, Budapest
  - Site Reference ID/Investigator# 54277, Győr
  - Site Reference ID/Investigator# 54275, Zalaegerszeg - Pozva
- Site Reference ID/Investigator# 54272, Udine, Italy
- Site Reference ID/Investigator# 54293, Amsterdam, Netherlands
- Poland (2):
  - Site Reference ID/Investigator# 54265, Gdansk
  - Site Reference ID/Investigator# 54266, Katowice
- Spain (2):
  - Site Reference ID/Investigator# 54280, Madrid
  - Site Reference ID/Investigator# 54264, Santiago de Compostela
- Site Reference ID/Investigator# 54271, Liverpool, United Kingdom